CLINICAL TRIAL: NCT03480737
Title: Intermittent Theta Burst Stimulation for Working Memory Deficits in Adolescents With ADHD
Brief Title: Brain Stimulation for Working Memory Deficits in Adolescents With ADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bradley Hospital (Other)
Collaborators: Thrasher Research Fund (Other); Rhode Island Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: BradleyH
Record Dates: First submitted 2018-03-12; First posted 2018-03-29 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: ADHD With Working Memory Deficits

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- 10 Hz rTMS (Experimental)
  Interventions: Device: Magstim Super Rapid2 stimulator, 10 Hz condition
- Sham rTMS (Sham Comparator)
  Interventions: Device: Magstim Super Rapid2 stimulator, Sham condition
- iTBS rTMS (Experimental)
  Interventions: Device: Magstim Super Rapid2 stimulator, iTBS condition

INTERVENTIONS:
Device: Magstim Super Rapid2 stimulator, 10 Hz condition — 10 Hz (2,000 pulses) at left DLPFC
  Arms: 10 Hz rTMS
Device: Magstim Super Rapid2 stimulator, Sham condition — sham
  Arms: Sham rTMS
Device: Magstim Super Rapid2 stimulator, iTBS condition — 50 Hz, iTBS (600 pulses) at left DLPFC
  Arms: iTBS rTMS

SUMMARY:
Working memory (WM) is the foundational cognitive control process of holding information 'in mind' to execute goal-directed behaviors. WM deficits are an established component of ADHD. Despite being one of the strongest predictors of poor clinical and functional outcomes in pediatric mental health, there remains a dearth of available treatments for WM deficits.

Non-invasive brain stimulation hold tremendous promise in transforming psychiatry, as it takes a "brain-first" approach to treatment. The dorsolateral prefrontal cortex (DLPFC) is the known structural foundation of WM, and the interaction between slow and fast brain waves (i.e., "theta-gamma coupling [TGC]") is a neural, functional foundation of WM. Thus, the DLPFC and TGC are potential brain-based targets for the modulation of WM with brain stimulation. Intermittent theta burst stimulation (iTBS) is a novel paradigm that applies a three-minute dose of stimulation to the DLPFC at an intensity that directly mimics TGC dynamics.

The objective of this study is to test whether iTBS can enhance dysfunctional brain activity that causes working memory deficits. iTBS will be tested compared to standard or traditional transcranial magnetic stimulation (TMS), called 10 Hz TMS. It will also be compared to sham or fake TMS. Each participant receives a single session of each of these types of TMS. EEG will record neural activity during a working memory test immediately before and after each TMS session. If this study shows TMS can enhance dysfunctional brain activity, the next step will be to conduct a clinical trial to test if TMS can lead to a sustained, positive effect on working memory deficits.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to provide assent and have parent provide parental permission
2. English fluency
3. 13-17 years
4. List Sorting Test (NIH Toolbox) performance: Greater than 1.0 standard deviation (SD) below normative mean
5. Parent rating on BRIEF-2 Working Memory: Greater than 1.0 SD above normative mean
6. IQ > 80
7. Clinical diagnosis of attention deficit hyperactivity disorder (ADHD): predominantly inattentive type, predominantly hyperactive/impulsive type, combined type, or unspecified type. Diagnostic criteria will be confirmed with NICHQ Vanderbilt Assessment Scales-Parent.

Exclusion Criteria:

Participants will be screened to exclude individuals with neurological or medical conditions that might confound the results, as well as to exclude participants in whom rTMS might result in increased risk of side effects or complications. Common TMS contraindications include metallic hardware in the body, cardiac pacemaker, patients with an implanted medication pumps or an intracardiac line, or prescription of medications known to lower seizure threshold. This accounts for the majority of the exclusion criteria listed:

1. Intracranial pathology from a known genetic disorder (e.g., NF1, tuberous sclerosis) or from acquired neurologic disease (e.g. stroke, tumor), cerebral palsy, history of severe head injury, or significant dysmorphology
2. History of fainting spells of unknown or undetermined etiology that might constitute seizures
3. History of seizures, diagnosis of epilepsy, or immediate (1st degree relative) family history epilepsy
4. Any progressive (e.g., neurodegenerative) neurological disorder
5. Chronic (particularly) uncontrolled medical conditions that may cause a medical emergency in case of a provoked seizure (cardiac malformation, cardiac dysrhythmia, asthma, etc.)
6. Contraindicated metal implants in the head, brain or spinal cord (excluding dental implants or fillings)
7. Pacemaker
8. Implanted medication pump
9. Vagal nerve stimulator
10. Deep brain stimulator
11. TENS unit (unless removed completely for the study)
12. Ventriculo-peritoneal shunt
13. Signs of increased intracranial pressure
14. Intracranial lesion (including incidental finding on MRI)
15. History of head injury resulting in prolonged loss of consciousness
16. Substance abuse or dependence within past six months (i.e., DSM-5 substance use disorder criteria met)
17. Chronic treatment with prescription medications that decrease cortical seizure threshold

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Compared to sham and 10 Hz, iTBS will enhance theta-gamma coupling during working memory demands | Within 24 hours

SECONDARY OUTCOMES:
Compared to sham and 10 Hz, iTBS will improve working memory test performance | Within 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Brian Kavanaugh, PsyD, Principal Investigator — E. P. Bradley Hospital/Alpert Medical School of Brown University
Locations (1):
- E. P. Bradley Hospital, East Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Undecided